CLINICAL TRIAL: NCT01938560
Title: REMS Prescriber and Pharmacist Understanding of the Risk of Urinary Retention With POTIGA™
Brief Title: REMS Retigabine Study
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 116490; WEUKBRE5993 (Other: GSK)
Record Dates: First submitted 2013-09-05; First posted 2013-09-10 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Physicians: Retigabine Physicians (e.g. neurologists/epileptologists/neurosurgeons) who have prescribed retigabine at least once in the last 12 months.
  Interventions: Other: Survey Responses
- Pharmacists: Pharmacists who have dispensed an anti-epileptic drug (AED) at least once in the last 3 months.
  Interventions: Other: Survey Responses

INTERVENTIONS:
Other: Survey Responses — Subject understanding of the risk of urinary retention and the symptoms of acute urinary retention associated with retigabine will be assessed using the survey instrument.

SUMMARY:
As part of a post-marketing commitment, GSK will conduct a survey of prescribers' and pharmacists' understanding of the risk of urinary retention with retigabine products. This is to address the effectiveness of the Risk Evaluation and Mitigation Strategy (REMS) as outlined in the REMS approved by the FDA on 10th June 2011. The objectives of this survey are to assess prescribers' and pharmacists' understanding of the risk of urinary retention and the symptoms of acute urinary retention potentially associated with retigabine use as evaluated by a survey instrument.

This is a cross-sectional study of approximately 200 physicians (e.g. neurologists/epileptologists/neurosurgeons) who have prescribed retigabine at least once in the last 12 months, and 200 pharmacists who have dispensed an anti-epileptic drug (AED) at least once in the last 3 months. The primary outcome of the survey is the proportion of physicians and pharmacists providing correct responses to a series of questions concerning the risk of urinary retention and the symptoms of acute urinary retention that may be associated with retigabine. The risks captured will be those described in the retigabine Dear Healthcare Provider (DHCP) letters, specifically risks of urinary retention.

DETAILED DESCRIPTION:
POTIGA is a trademark of Valeant Pharmaceuticals North America, used by GlaxoSmithKline under license.

ELIGIBILITY:
Inclusion Criteria:

* Able to read, speak, and understand English.
* Willing to take the online survey or have the survey administered via a telephone interview, including electronically signing a Confidentiality & Consent agreement and completing all study protocol-specified procedures.
* Prescribed retigabine within the past 12 months (prescribing physicians)
* Filled a prescription for at least one AED within the previous three months (pharmacists).

Exclusion Criteria:

* Physicians or pharmacists meeting any of the following criteria will not be eligible to take the survey:
* The physician or pharmacist is currently employed by, or is a representative of any of the following:
* A pharmaceutical company or manufacturer of medicines or healthcare products.
* Contributor/editor to published guideline committees for epilepsy or UR.
* The physician or pharmacist has a visual impairment that would prevent him or her from being able to read independently.
* The physician or pharmacist participated in the Pilot REMS study for retigabine.
* The physician or pharmacist is an employee of GSK or Concentrics Research.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 200 physicians (e.g. neurologists/epileptologists/neurosurgeons) who have prescribed retigabine at least once in the last 12 months, and 200 pharmacists who have dispensed an anti-epileptic drug (AED) at least once in the last 3 months.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2013-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
The proportion of physicians and pharmacists providing correct responses to a series of questions concerning the risk of urinary retention and the symptoms of acute urinary retention that may be associated with retigabine. | 12 months
  The outcome is a survey response by physicians and pharmacists so is not related to the drug exposure.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline